CLINICAL TRIAL: NCT03813563
Title: Lactated Ringer's and PlasmaLyte in Critically Ill Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, Clinical Professor, West China Hospital
Other Study IDs: RL vs Plalyte
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mix group: Patients who used two balanced salt solutions during icu stay
  Interventions: Drug: RL; Drug: PLA
- RL group: Patients who have only used lactated Ringer's during icu stay
  Interventions: Drug: RL
- PLA group: Patients who have only used PlasmaLyte during icu stay
  Interventions: Drug: PLA

INTERVENTIONS:
Drug: RL — lactated Ringer's
  Groups: Mix group; RL group
Drug: PLA — PlasmaLyte
  Groups: Mix group; PLA group

SUMMARY:
In recent years, there has been a large amount of literature reports that normal saline can increase the incidence of renal injury in critically ill patients compared with balanced salt solution.However, no studies have compared the effects of different types of balanced salt solutions on the incidence of renal injury.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to ICU

Exclusion Criteria:

* Patients <18 year old when admission
* Patients who stay less than 24 hours in ICU
* Patients who do not sufficient data for further analysis
* Readmission patients during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU admissions
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute kidney injury | from admission to 28 days
  The incidence of acute kidney injury

SECONDARY OUTCOMES:
the incidency of CRRT events | from admission to 28 days
  the incidency of CRRT events
the ventilation free days | from admission to 28 days
  the ventilation free days
the vasopressure free days | from admission to 28 days
  the vasopressure free days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical care medicine of West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided